CLINICAL TRIAL: NCT01812707
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study Evaluating the Efficacy and Safety of Three Doses of SAR236553 (REGN727) Over 12 Weeks in Patients With Primary Hypercholesterolemia and LDL-cholesterol ≥100 mg/dL (≥2.59 mmol/L) on Ongoing Stable Atorvastatin Therapy
Brief Title: Efficacy and Safety Evaluation of Alirocumab (SAR236553/REGN727) in Patients With Primary Hypercholesterolemia on Stable Atorvastatin Therapy in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI12361; U1111-1134-4749 (Other: UTN)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2015-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo (for alirocumab) every 2 weeks (Q2W) for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Placebo (for alirocumab); Drug: Atorvastatin
- Alirocumab 50 mg Q2W (Experimental): Alirocumab 50 mg Q2W for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin
- Alirocumab 75 mg Q2W (Experimental): Alirocumab 75 mg Q2W for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin
- Alirocumab 150 mg Q2W (Placebo Comparator): Alirocumab 150 mg Q2W for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin

INTERVENTIONS:
Drug: Alirocumab — Two SC injections in the abdomen only
  Other Names: SAR236553; RGEN727
  Arms: Alirocumab 150 mg Q2W; Alirocumab 50 mg Q2W; Alirocumab 75 mg Q2W
Drug: Placebo (for alirocumab) — Two subcutaneous (SC) injections in the abdomen only
  Route of administration: subcutaneous injection (1 mL) in the abdomen
  Arms: Placebo
Drug: Atorvastatin — Orally once daily at a stable dose of 5 to 20 mg as background therapy
  Route of administration: oral administration in the evening

SUMMARY:
Alirocumab (SAR236553/REGN727) is a fully human monoclonal antibody that binds proprotein convertase subtilisin/kexin type 9 (PCSK9).

Primary Objective of the study:

To evaluate the effect of alirocumab on low-density lipoprotein cholesterol (LDL-C) levels after 12 weeks of treatment in comparison with placebo in participants with LDL-C ≥100 mg/dL (≥2.59 mmol/L) on ongoing stable atorvastatin therapy.

Secondary Objectives:

* To evaluate the effects of alirocumab on other lipid levels after 12 weeks of treatment in comparison with placebo
* To evaluate the safety and tolerability of alirocumab
* To evaluate the development of anti-alirocumab antibodies
* To evaluate the pharmacokinetics of alirocumab

DETAILED DESCRIPTION:
The duration of study participation depended on the status of the participant at screening: 21 to 27 weeks including a screening/run-in period of 1 to 7 weeks, a double-blind treatment period of 12 weeks, followed by an 8-week follow-up period.

ELIGIBILITY:
Inclusion criteria :

- Participants with primary hypercholesterolemia treated with atorvastatin at stable dose of 5-20 mg for at least 6 weeks prior to screening and likely to have LDL-C ≥100 mg/dL (≥2.59 mmol/L) at the screening visit.

OR

- Participants with primary hypercholesterolemia who were receiving a lipid-lowering treatment other than atorvastatin, or who were not at stable dose of atorvastatin 5-20 mg for at least 6 weeks prior to screening if they were likely to have LDL-C ≥100 mg/dL (≥2.59 mmol/L) after a 6-week run-in treatment period on atorvastatin therapy.

Exclusion criteria:

1. LDL-C <100 mg/dL (<2.59 mmol/L)

   * at screening visit for participants who were being treated with stable dose of atorvastatin 5-20 mg for at least 6 weeks prior to screening OR
   * at the end of the 6-week run-in period on atorvastatin for participants receiving a lipid lowering treatment other than atorvastatin, or not at stable dose of atorvastatin 5-20 mg for at least 6 weeks prior to screening
2. Participants with type 1 diabetes
3. Participants with type 2 diabetes treated with insulin, or without, and considered poorly controlled at screening.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Japan (4):
  - Investigational Site Number 392002, Koganeishi
  - Investigational Site Number 392001, Shinjuku-Ku
  - Investigational Site Number 392003, Suita-Shi
  - Investigational Site Number 392004, Suita-Shi

REFERENCES:
- [Result] Teramoto T, Kobayashi M, Uno K, Takagi Y, Matsuoka O, Sugimoto M, Inoue S, Minami F, Baccara-Dinet MT. Efficacy and Safety of Alirocumab in Japanese Subjects (Phase 1 and 2 Studies). Am J Cardiol. 2016 Jul 1;118(1):56-63. doi: 10.1016/j.amjcard.2016.04.011. Epub 2016 Apr 21. PMID 27184170
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 centers in Japan. Overall, 162 participants were screened between March 2013 and August 2013, 62 of whom were run-in/screen failures, mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to atorvastatin dose. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:1:1:1 ratio after confirmation of selection criteria. 100 participants were randomized.
Period: Overall Study
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Started | 25 | 25 | 25 | 25
Treated | 25 | 25 | 25 | 25
Completed | 23 | 25 | 25 | 23
Not Completed | 2 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Poor compliance to protocol | 1 | 0 | 0 | 0
Not completed — Consent withdrawn by participant | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population.
Groups:
- Placebo: Placebo (for alirocumab) Q2W for 12-weeks in combination with atorvastatin stable dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.2) | 57.8 (12.3) | 56.3 (12.0) | 58.2 (8.8) | 57.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 12 | 16 | 55
  Male | 14 | 9 | 13 | 9 | 45
Low-Density Lipoprotein Cholesterol (LDL-C) in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 3.13 (0.55) | 3.16 (0.43) | 3.13 (0.43) | 3.12 (0.42) | 3.14 (0.45)
LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] | 121.0 (21.1) | 122.2 (16.6) | 120.9 (16.7) | 120.5 (16.2) | 121.2 (17.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Calculated LDL-C values were obtained using the Friedewald formula. Baseline adjusted least squares (LS) means and standard errors were estimated using an analysis of covariance (ANCOVA) model including available post-baseline data on treatment from first investigational product (IP) injection up to 21 days after last IP injection (on-treatment analysis). Missing Week 12 data were imputed by last observation carried forward [LOCF] method.
Time Frame: Baseline to Week 12 (LOCF)
Population: Modified Intent-To-Treat (mITT) population included all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 25 | 25 | 25 | 25
percent change | -2.7 (3.1) | -54.8 (3.1) | -62.3 (3.1) | -71.7 (3.1)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 150 mg Q2W; Each treatment group was compared to placebo using ANCOVA-derived contrasts. A hierarchical testing procedure was applied to ensure strong control of overall Type-I error rate at 0.05 level. Order was following: 1. Alirocumab 150 mg Q2W versus placebo 2. Alirocumab 75 mg Q2W versus placebo 3. Alirocumab 50 mg Q2W versus placebo Testing continued only when high-order test was statistically significant at 5% level; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤0.05
Statistical Analysis 2: Comparison: Placebo vs Alirocumab 75 mg Q2W; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤0.05
Statistical Analysis 3: Comparison: Placebo vs Alirocumab 50 mg Q2W; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤0.05

2. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C (mmol/L) at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: Baseline to Week 12 (LOCF)
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 25 | 25 | 25 | 25
mmol/L | -0.1 (0.1) | -1.7 (0.1) | -1.9 (0.1) | -2.2 (0.1)

3. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C (mg/dL) at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: Baseline to Week 12 (LOCF)
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 25 | 25 | 25 | 25
mg/dL | -5.0 (3.6) | -67.1 (3.6) | -74.6 (3.6) | -85.8 (3.6)

4. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <100 mg/dL (2.59 mmol/L) and < 70 mg/dL (1.81 mmol/L) at Week 12 - On-Treatment Analysis
Time Frame: Week 12 (LOCF)
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 25 | 25 | 25 | 25
percentage of participants
  LDL-C <100 mg/dL (2.59 mmol/L) | 8.0 | 100.0 | 100.0 | 100.0
  LDL-C < 70 mg/dL (1.81 mmol/L) | 0.0 | 84.0 | 84.0 | 88.0

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol, High-Density Lipoprotein Cholesterol (HDL-C), Non-HDL-C, and Apolipoprotein B (Apo-B) at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: Baseline to Week 12 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post baseline on-treatment value of lipid parameters analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 25 | 25 | 25 | 25
percent change
  Total Cholesterol | -1.2 (2.1) | -31.9 (2.1) | -36.3 (2.1) | -41.4 (2.1)
  HDL-C | -0.2 (2.0) | 5.1 (2.0) | 5.0 (2.0) | 3.2 (2.1)
  Non-HDL-C | -0.9 (2.9) | -46.3 (2.9) | -53.1 (2.9) | -62.2 (2.9)
  Apo-B | -2.3 (3.3) | -43.5 (3.3) | -48.6 (3.3) | -60.0 (3.3)

6. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides and Lipoprotein (a) at Week 12 - On-Treatment Analysis
Description: Since the assumptions of normal distribution and equality of variances were not verified for the lipid parameters, percent changes were expressed as median (inter-quartile range).
Time Frame: Baseline to Week 12 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post baseline on-treatment value of Fasting Triglycerides and Lipoprotein (a) analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 25 | 25 | 25 | 25
percent change
  Fasting Triglycerides | 1.3 [-13.1 to 22.5] | -21.1 [-28.2 to 4.2] | -10.7 [-25.0 to 6.5] | -15.0 [-24.1 to 0.0]
  Lipoprotein (a) | -3.7 [-26.2 to 8.4] | -35.6 [-52.5 to -7.5] | -40.2 [-62.9 to -27.4] | -43.3 [-69.4 to -14.2]

7. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein B/Apolipoprotein A-1 (ApoB/ApoA-1) Ratio at Week 12 - On-Treatment Analysis
Description: Adjusted LS mean and standard errors were estimated using the same ANCOVA as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post baseline on-treatment value of ApoB/ApoA-1 ratio analyzed.
Measure: Least Squares Mean (Standard Error); unit: ratio
Groups:
- Placebo: Placebo (for alirocumab) Q2W for 12 weeks in combination with atorvastatin stable dose.
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 25 | 25 | 25 | 25
ratio | 0.02 (0.02) | -0.30 (0.02) | -0.32 (0.02) | -0.38 (0.02)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 20) regardless of seriousness or relationship to investigational medicinal product (IMP).
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment emergent period' (the time from the first dose to the last dose of IMP + 70 days). Safety population: participants who received at least one dose or partial dose of IMP.
Groups:
- Placebo: Placebo Q2W for 12 weeks in combination with atorvastatin stable dose.
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 75 mg Q2W | Alirocumab 150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25 | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 5/25 | 11/25 | 8/25 | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | Alirocumab 50 mg Q2W (N=25) | Alirocumab 75 mg Q2W (N=25) | Alirocumab 150 mg Q2W (N=25)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | Alirocumab 50 mg Q2W (N=25) | Alirocumab 75 mg Q2W (N=25) | Alirocumab 150 mg Q2W (N=25)
Nasopharyngitis (Infections and infestations) | 2 | 6 | 6 | 4
Cystitis (Infections and infestations) | 1 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Injection site reaction (General disorders) | 1 | 3 | 2 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.